CLINICAL TRIAL: NCT04051801
Title: Multiple Ascending Dose Phase I Study of the M1 Positive Allosteric Modulator VU0467319
Brief Title: Multiple Ascending Dose Putative Cognitive Enhancer VU319
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Further development has been outlicensed to Acadia Pharmaceuticals
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Paul Newhouse, MD, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190919
Record Dates: First submitted 2019-07-19; First posted 2019-08-09 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple-blind safety study. The pharmacist is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation of VU319 - Dose 1 (Experimental)
  Interventions: Drug: Dose Escalation of VU319; Drug: Dose Escalation of Placebo
- Dose Escalation of Placebo - Dose 1 (Placebo Comparator)
  Interventions: Drug: Dose Escalation of VU319; Drug: Dose Escalation of Placebo
- Dose Escalation of VU319 - Dose 2 (Experimental)
  Interventions: Drug: Dose Escalation of VU319; Drug: Dose Escalation of Placebo
- Dose Escalation of Placebo - Dose 2 (Placebo Comparator)
  Interventions: Drug: Dose Escalation of VU319; Drug: Dose Escalation of Placebo
- Dose Escalation of VU319 - Dose 3 (Experimental)
  Interventions: Drug: Dose Escalation of VU319; Drug: Dose Escalation of Placebo
- Dose Escalation of Placebo - Dose 3 (Placebo Comparator)
  Interventions: Drug: Dose Escalation of VU319; Drug: Dose Escalation of Placebo

INTERVENTIONS:
Drug: Dose Escalation of VU319 — dose levels of the cohorts will be increased step wise
Drug: Dose Escalation of Placebo — dose levels of the cohorts will be increased step wise

SUMMARY:
This is a safety study of the molecule VU319 to ascertain pharmacokinetic and pharmacodynamic data and test cognitive enhancement in healthy volunteers.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a chronic and irreversible neurodegenerative disease characterized by the deterioration of memory and other cognitive functions, progressive impairments in normal daily living, and severe neuropsychiatric symptoms and behavioral disturbances. Currently, there is no available prevention or cure for AD. Therapeutic strategies for the cognitive impairments in AD involve only symptomatic treatments, primarily through enhancement of cholinergic neurotransmission using AChEIs.

Primary objectives To establish the safety and tolerability of multiple dose (up to VU319 steady state) VU319 administration in healthy volunteers To establish the maximum tolerated dose of multiple dose (up to VU319 steady state) VU319 administration in healthy volunteers To characterize the plasma pharmacokinetics and urinary excretion of VU319 and metabolite after single dose oral administration in healthy volunteers Secondary objectives To establish the effect of food on the bioavailability and pharmacokinetic parameters of VU319 in healthy volunteers Exploratory Objectives To gain preliminary evidence that tolerable doses of VU319 engage central M1 receptors by 1) altering/enhancing cognitive performance, and 2) enhancing cortical event related potentials (ERP) as a measure of increased cognitive function in healthy volunteers

This will be a double blind, randomized, placebo controlled, and sequential dose escalation in male or female healthy volunteers. Gender will be balanced to the extent possible. Volunteers will receive oral VU319 multiple dose administration in the fasted state. Subjects meeting entry criteria will be enrolled in successive dose escalating cohorts of 8 subjects each (2 placebo and 6 active drug per dose level). The dose levels will be tested sequentially until the Maximum Tolerated Dose (MTD) is reached, or saturation of exposure occurs, or sustained VU319 plasma level above the safe daily exposure determined from animal toxicokinetic studies is achieved.

Clinical safety endpoints include adverse event and symptoms data, vital signs (HR, BP, Respiratory Rate, body weight), 12-lead ECG changes, and laboratory safety assessments (hematology, plasma biochemistry, coagulation, urinalysis).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 through 55 years, inclusive.
2. Body mass index 18 through 32 kg/m2
3. Determined as healthy based on screening medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG without clinically significant abnormalities. QTc interval with Fridericia's correction method recorded on screening and predose must be less than 450 msec for male and less than 470 in females.
4. Clinical laboratory test result without clinically significant abnormalities at screening and at admission.
5. Negative tests for Hepatitis B surface antigen, hepatitis C virus antibodies and human immunodeficiency virus (HIV-1 or HIV-2) antibody at screening.
6. Nonsmokers (use of any nicotine containing product) or ex-smokers (have ceased smoking for at least 6 months and do not use any drug for smoking cessation).
7. Negative screen for drugs of abuse at screening and admission.
8. Negative screen for alcohol at admission.
9. For Women: Must have no child-bearing potential by reason of a sterilization procedure or at least 1 year post-menopausal (i.e. 12 months without menstrual period), or menopause confirmed with follicle-stimulating hormone level of > 30 IU/L at screening.
10. For Men: Must be infertile (at least 3-months post-vasectomy), or truly abstinent of heterosexual intercourse, or heterosexual partner is not of child-bearing potential or must agree to use an effective method of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository) through the study and for 28 days after last dose of study drug.
11. Able and willing to be available for the duration of the study.
12. Willing and able to give written informed consent to participate.
13. Able to understand and comply with protocol instructions.
14. Agrees not to receive any vaccination within 21 days prior to admission and through Day 7 after final discharge.
15. Agrees not to use nonprescription drugs, including vitamins, antacids, and herbal and dietary supplements within 7 days prior to admission and through 7 days after final discharge. Acetaminophen may be used at doses of ≤ 1 g/day, and ibuprofen may be used at doses of ≤ 1.2 g/day.
16. Agrees not to use nicotine-containing products from screening through 48 hours after discharge.
17. Agrees not to consume alcohol for the 72 hours prior to admission and through 48 hours after discharge.
18. Agrees not to eat grapefruit or drink grapefruit juice within 7 days prior to admission and through 24 hours after discharge.
19. Agrees to not drink caffeinated drinks from 72 hours prior to admission through discharge.
20. Agrees not to eat or drink (except water) for 8 hours before and 4 hour after dosing for all MAD cohort subjects.

Exclusion Criteria:

1. Individuals with significant previous or ongoing disease or disorder, based on history, physical exam, ECG, and laboratory tests, including for example: Cardiovascular diseases; hypertension; cancer or neoplasia; diabetes; hepatic, endocrine, metabolic, respiratory, renal, gastrointestinal (except appendectomy), dermatological or hematological disorders, Axis I or II psychiatric, substance use, or cognitive disorders.
2. Clinically significant infection or inflammation at time of admission.
3. Clinically significant abnormalities upon physical/neurological exam at screening.
4. Acute gastrointestinal symptoms (e.g. nausea, vomiting, diarrhea) at admission
5. History of treatment from a physician or counselor for abuse or misuse of alcohol, non-prescription drugs, medicinal drugs or other substance abuse.
6. Any current or previous use of Class A drugs such as illicit opiate use, cocaine, ecstasy, LSD, and amphetamines (Class B). Volunteers that admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs-of-abuse test at screening and admission and have been abstinent for at least 3 months.
7. An alcoholic intake greater than 21 units per week or unwillingness to stop alcohol consumption for the duration of the study. Note: 1 unit = 8 g ethanol (250 mL of beer, 1 glass wine [100 mL], 1 measure spirits [30 mL]).
8. Use of medication (including OTC and oral contraceptive agents) within 14 days of admission that may affect the safety of the subject or any study assessment, in the opinion of the investigator.
9. Use of prescribed centrally active or psychoactive agents within 28 days prior to admission.
10. Requirement for any medication that would need to be continued during the study.
11. Use of any investigational medication within 3 months prior to the start of this study or scheduled to receive an investigational drug during the course of this study.
12. Have participated in more than 2 clinical trials involving research medication use within the 12 months prior to screening.
13. History of blood donation in the 2 months prior to admission.
14. History of severe allergies or multiple adverse drug reactions.
15. Any condition, which compromises ability to give informed consent or to communicate with the investigator as required for the completion of this study.
16. The subject has been previously enrolled in the MAD study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Changes in adverse events frequency from Baseline to 144 hours post last drug administration
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Cognitive Battery - Critical Flicker Fusion (CFF) | Baseline, 1 hours post last drug administration
  The Critical Flicker Fusion (CFF) task will be used as a test of vigilance. The primary dependent measures are ascending and descending fusion frequency (Hz).
Cognitive Battery - Choice Reaction Time (CRT) | Baseline, 1 hours post last drug administration
  The Choice Reaction Time (CRT) task from the Milford Test Battery will be used to examine psychomotor functions. The dependent measures are the median total reaction time (RT), and its subcomponents of recognition RT, motor RT.
Cognitive Battery - Spatial Selective Attention (Posner Task) | Baseline, 1 hours post last drug administration
  This task measures response speed corresponding to a validly and invalidly cued stimulus. The cue will be valid 57% of the time, and for the other 43% will be equiprobable as an invalid cue, a neutral cue showing pointing to both sides, or a no cue condition. The two outcome measures will be difference scores between the cues. The first is the alerting effect (neutral - no cue trials). The second is the reorienting effect (valid - invalid trials).
Cognitive Battery - Continuous Performance Test (Conners) | Baseline, 1 hours post last drug administration
  The Conners Continuous Performance Task (CPT) will be used to measure sustained attention. The dependent measures are omission and commission errors, hit reaction time, hit RT standard error (SE).
Cognitive Battery - Working Memory (N-Back Test) | Baseline, 1 hours post last drug administration
  The N-Back Test will be used as a test of verbal working memory. The dependent measures are sensitivity (d') and bias (C) across load conditions (0-3 back).
Cognitive Battery - The Selective Reminding Task (SRT) | Baseline, 1 hours post last drug administration
  The Selective Reminding Task (SRT) is a multi-trial verbal list-learning task allowing the examination of acquisition, encoding and retrieval. This standard test has been widely used in studies of cognitive impairment and offers measures of storage into and retrieval from both short term and long-term memory and intrusion errors. The dependent measures are immediate total (8 trials) word recall, recall failure, recall consistency and delayed recall.
Cognitive Battery - Trail Making Task | Baseline, 1 hours post last drug administration
  The Trail Making Task is a neuropsychological test of visual attention and task switching. The dependent measurement will be the difference in completion time between Trails B and Trails A.
Event-Related Potentials- Incidental Memory Tasks | Baseline, 2.5 hours post last drug administration
  Change in late positive potential (P300-600) amplitude over frontal, central, and parietal midline locations (Fz, Cz, Pz) for repeated vs novel stimuli.
Event-Related Potentials- Auditory and Visual Oddball Tasks | Baseline, 2.5 hours post last drug administration
  Change in P300 amplitude over frontal, central, and parietal midline locations (Fz, Cz, Pz) for target vs standard stimuli.
Quantitative EEG | Baseline, 2.5 hours post last drug administration
  A passive 3 minutes resting-EEG paradigm, with two blocks, one with eyes closed, the other with eyes open. The dependent variable for this paradigm will be changes in power of frequency bands from 2-30 Hz between baseline and post-dose testing sessions.
Behavioral Measure - Profile of Mood State (POMS) | Baseline, 1 hours post last drug administration
  The Profile of Mood States (POMS) measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A five-point scale ranging from "not at all" to "extremely" is administered by experimenters to patients to assess their mood states.
Behavioral Measure - Brief Psychiatric Rating Scale (BPRS) | Baseline, 1 hours post last drug administration
  Brief Psychiatric Rating Scale (BPRS) assesses the level of 24 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. It is particularly useful in gauging the efficacy of treatment in patients who have moderate to severe psychoses. It is based on the clinician's observations of the patient's behavior. The rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe).
Behavioral Measure - Subject Visual Analogue Scale (SVAS) | Baseline, 1 hours post last drug administration
  Subject Visual Analog Scales (SVAS) will be used consisting of a series of items such as "drowsiness" or "psychomotor agitation" scored on 100 mm lines scored by the subject.
Behavioral Measure - Stanford Sleepiness Scale | Baseline, 0.5 hour pre each drug administration and 23.5 hour post last drug administration
  To collect a spectrum of sleepiness indicators across a day, the SSS is administered at two-hour intervals. The SSS uses the following numeric scale:
  1. Feeling active, vital, alert, and wide awake.
  2. Functioning at a high level but not at peak performance. Able to concentrate.
  3. Relaxed and awake, but not fully alert. Still responsive.
  4. Feeling a little foggy and let down.
  5. Foggy and beginning to lose track of things. Difficult to stay awake.
  6. Sleepy and prefer to lie down. Woozy.
  7. Almost in reverie and cannot stay awake. Sleep onset is imminent.
Behavioral Measure - Physical Symptom Checklist | Baseline, 0.5 hour pre each drug administration and 23.5 hour post last drug administration
  A checklist of 22 physical symptoms. Each item is rated 1 to 4, with 1 being none and 4 being severe. Total score range from 22 to 88.
Actigraphy | Day-1 (Baseline) to Day 8 (23.5 hour post last drug administration)
  Starting at day -1, each subject will receive a wearable motion-based actigraphy device for assessing sleep (sleep duration and patterns of deep and light sleep stages) and biometrics. The device incorporates clinical-grade photoplethysmography (PPG) technology to capture physiological biometric data, including heart rate (HR), heart rate variability (HRV), respiratory rate(RR), and blood oxygen saturation (SPO2).
Behavioral Measure-Suicide Behavior Questionnaire (SBQ-R) | Day 8 (23.5 hour post last drug administration), Day 12(144 hours post last drug administration)
  It consists of four questions. Each of the four questions addresses a specific risk factor: the first concerns presence of suicidal thoughts and attempts, the second concerns frequency of suicidal thoughts, the third concerns the threat level of suicidal attempts, and the fourth concerns likelihood of future suicidal attempts. The first item has often been used on its own in order to assign individuals to a suicidal and a non-suicidal control group for studies. A total score of 7 and higher in the general population and a total score of 8 and higher in patients with psychiatric disorders indicates significant risk of suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Newhouse, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States